CLINICAL TRIAL: NCT00784550
Title: A Randomized, Double-Blind, Parallel-Group, 24-Week Study to Evaluate the Efficacy and Safety of ADVAIR DISKUS (Fluticasone Propionate/Salmeterol Combination Product 250/50mcg Inhalation Powder) BID Plus Spiriva HandiHaler (Tiotropium Bromide Inhalation Powder 18mcg) QD Versus Spiriva QD Plus Placebo DISKUS BID in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 24-Week Study to Evaluate the Safety and Efficacy of ADVAIR DISKUS® Inhaler 250/50mcg Plus SPIRIVA HANDIHALER® Inhaler Versus SPIRIVA HANDIHALER® Inhaler Plus Placebo DISKUS® Inhaler in Subjects With Chronic Obstructive Pulmonary Disease (COPD).
Acronym: ADC111114
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111114
Record Dates: First submitted 2008-10-31; First posted 2008-11-04 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Spirometry; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADVAIR DISKUS® inhlaer Plus SPIRIVA® HANDIHALER® inhaler (Experimental): Fluticasone Propionate/Salmeterol Combination Product 250/50mcg BID Plus Tiotropium Bromide 18 mcg QD
  Interventions: Drug: Fluticasone Propionate/Salmeterol
- SPIRIVA® HANDIHALER® inhaler (Active Comparator): Tiotropium Bromide 18mcg QD plus Placebo DISKUS BID
  Interventions: Drug: Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium Bromide — Long-acting muscarinic antagonist
  Arms: SPIRIVA® HANDIHALER® inhaler
Drug: Fluticasone Propionate/Salmeterol — Inhaled corticosteroid plus long-acting bronchodilator
  Arms: ADVAIR DISKUS® inhlaer Plus SPIRIVA® HANDIHALER® inhaler

SUMMARY:
The purpose of the study is to determine the efficacy and safety of the combination of ADVAIR DISKUS® 250/50mcg (FLUTICASONE PROPIONATE/SALMETEROL COMBINATION PRODUCT) plus SPIRIVA® HANDIHALER® inhaler 18mcg (TIOTROPIUM) compared to SPIRIVA® HANDIHALER® inhaler 18mcg (TIOTROPIUM) in patients with COPD.

SPIRIVA® and HANDIHALER® are trade marks of Boehringer Ingelheim Pharma GmbH & Co. KG.

ADVAIR DISKUS® are registered trademarks of the GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis
* At least 10 pack year smoking history
* Post-albuterol FEV1 greater than or equal to 40% to less than or equal to 80% of predicted normal
* An FEV1/FVC ratio of less than or equal to 0.70

Exclusion Criteria:

* Current diagnosis of asthma
* Other respiratory disorder other than COPD
* Abnormal and clinical significant ECG
* Chest x-ray clinically significant abnormality not believed to be due to COPD
* Body Mass Index of greater than or equal to 40/kg/m2
* Use of Long Term Oxygen Therapy
* Lung resection surgery
* Women pregnant or lactating at Visit 1
* Previously diagnosed cancer unless in complete remission for 2 years at Visit 1

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (34):
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Naranja, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Gillespie, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Olathe, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Milan, Tennessee
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Hanania NA, Crater GD, Morris AN, Emmett AH, O'Dell DM, Niewoehner DE. Benefits of adding fluticasone propionate/salmeterol to tiotropium in moderate to severe COPD. Respir Med. 2012 Jan;106(1):91-101. doi: 10.1016/j.rmed.2011.09.002. Epub 2011 Oct 29. PMID 22040533
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111114 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- FSC + Tio: Open-label tiotropium (Tio) 18 micrograms (mcg) once-daily (QD) plus double-blind Fluticasone Propionate/Salmeterol Combination (FSC) 250/50 mcg twice daily (BID)
- Tiotropium: Open-label Tio 18 mcg QD plus double-blind matching placebo DISKUS BID
Period: Overall Study
Arm/Group | FSC + Tio | Tiotropium
Started | 173 | 169
Completed | 137 | 127
Not Completed | 36 | 42
Not completed — Adverse Event | 12 | 10
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 10 | 10
Not completed — Lost to Follow-up | 8 | 5
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 4 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSC + Tio | Tiotropium | Total
Number analyzed (Participants) | 173 | 169 | 342
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (8.56) | 61.0 (9.41) | 61.2 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 96 | 182
  Male | 87 | 73 | 160
Race/Ethnicity, Customized [Number; unit: participants]
  White | 165 | 162 | 327
  African American/African Heritage | 7 | 7 | 14
  American Indian or Alaska Native | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in AM (Morning, Approximately 6-9 AM) Pre-dose Forced Expiratory Volume in One Second (FEV1) at Endpoint
Description: Change from baseline was calculated as the Endpoint (defined as the last recorded measure of AM pre-dose FEV1 for each participant) value minus the baseline value. FEV1 is defined as the amount of air expelled from the lungs in one second after a full inspiration and is a measure of pulmonary function.
Time Frame: Baseline and Endpoint (defined as the last recorded measure [taken up to Week 24] of AM pre-dose FEV1 for each participant)
Population: Intent-to-Treat (ITT) Population: all participants randomized to study drug
Measure: Mean (Standard Error); unit: milliliters (ml)
Arm/Group | FSC + Tio | Tiotropium
Number analyzed (Participants) | 173 | 169
milliliters (ml) | 101 (21.8) | -16 (20.4)
Statistical Analysis 1: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Mean Change From Baseline in 2 Hour Post-dose FEV1 at Endpoint
Description: Change from baseline was calculated as the Endpoint (defined as the last recorded measure of 2 hour post-dose FEV1 for each participant) value minus the baseline value. FEV1 is defined as the amount of air expelled from the lungs in one second after a full inspiration and is a measure of pulmonary function.
Time Frame: Baseline and Endpoint (defined as the last recorded measure [taken up to Week 24] of 2 hour post-dose FEV1 for each participant)
Population: ITT Population
Measure: Mean (Standard Error); unit: ml
Arm/Group | FSC + Tio | Tiotropium
Number analyzed (Participants) | 173 | 169
ml | 233 (23.1) | 77 (20.6)
Statistical Analysis 1: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Secondary Outcome: Mean Change From Baseline in AM (Morning, Approximately 6-9 AM) Pre-dose Forced Vital Capacity (FVC) at Endpoint
Description: Change from baseline was calculated as the Endpoint (defined as the last recorded measure of AM pre-dose FVC fore each participant) value minus the baseline value. FVC is defined as the amount of air that can forcibly be blown out after a full inspiration.
Time Frame: Baseline and Endpoint (defined as the last recorded measure [up to Week 24] of AM pre-dose FVC for each participant)
Population: ITT Population
Measure: Mean (Standard Error); unit: ml
Arm/Group | FSC + Tio | Tiotropium
Number analyzed (Participants) | 173 | 169
ml | 95 (32.7) | -28 (30.6)
Statistical Analysis 1: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p = 0.006, ANCOVA

4. Secondary Outcome: Mean Change From Baseline in 2 Hour Post-dose FVC at Endpoint
Description: Change from baseline was calculated as the Endpoint (defined as the last recorded measure of 2 hour post-dose FVC for each participant) value minus the baseline value. FVC is defined as the amount of air that can forcibly be blown out after a full inspiration (FVC).
Time Frame: Baseline and Endpoint (defined as the last recorded measure of 2 hour post-dose FVC [up to Week 24] for each participant)
Population: ITT Population
Measure: Mean (Standard Error); unit: ml
Arm/Group | FSC + Tio | Tiotropium
Number analyzed (Participants) | 173 | 169
ml | 265 (35.9) | 87 (31.2)
Statistical Analysis 1: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Mean Change From Baseline in AM (Morning, Approximately 6-9 AM) Pre-Dose Inspiratory Capacity (IC) at Endpoint
Description: Change from baseline was calculated as the Endpoint (defined as the last recorded measure of AM pre-dose IC for each participant) value minus the baseline value. IC is defined as the amount of air that can be inhaled after a normal expiration. IC is a measure of pulmonary function.
Time Frame: Baseline and Endpoint (defined as the last recorded measure of AM pre-dose IC [up to Week 24] for each participant)
Population: ITT Population
Measure: Mean (Standard Error); unit: ml
Arm/Group | FSC + Tio | Tiotropium
Number analyzed (Participants) | 173 | 169
ml | 107 (28.4) | -8 (28.1)
Statistical Analysis 1: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Mean Change From Baseline in Scores on the Chronic Respiratory Disease Questionnaire-Self-Administered Standardized (CRQ-SAS) at Endpoint
Description: The CRQ-SAS measures 4 domains of functioning of participants with COPD: mastery (amount of control the participant feels he/she has over COPD symptoms); fatigue (how tired the participant feels); emotional function (how anxious/depressed the participant feels); and dyspnea (how short of breath the participant feels during physical activities). Each domain is measured on a scale of 1-7 (1=maximum impairment; 7=no impairment). Each domain score is calculated separately.
Time Frame: Baseline and Endpoint (defined as the last recorded score [up to Week 24 or the early withdrawal visit] on each of the questions on this questionnaire)
Population: ITT Population
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | FSC + Tio | Tiotropium
Number analyzed (Participants) | 173 | 169
points on a scale
  Mastery | 0.28 (0.078) | 0.04 (0.090)
  Fatigue | 0.23 (0.094) | 0.17 (0.091)
  Emotional Function | 0.24 (0.072) | 0.16 (0.073)
  Dyspnea | 0.21 (0.091) | 0.19 (0.091)
Statistical Analysis 1: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p = 0.069, ANCOVA — Mastery domain
Statistical Analysis 2: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p = 0.470, ANCOVA — Fatigue domain
Statistical Analysis 3: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p = 0.394, ANCOVA — Emotional function domain
Statistical Analysis 4: Comparison: FSC + Tio vs Tiotropium; Test type: Superiority or Other; p = 0.879, ANCOVA; Dyspnea domain

ADVERSE EVENTS:
Description: The serious adverse events of finger amputation and shoulder amputation were actually coded to the system organ class of surgical and medical procedures.
Arm/Group | FSC + Tio | Tiotropium
Serious Adverse Events (participants affected / at risk) | 7/173 | 13/169
Other Adverse Events (participants affected / at risk) | 34/173 | 29/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC + Tio (N=173) | Tiotropium (N=169)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Ileus (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Gastric infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Finger amputation (Injury, poisoning and procedural complications) | 0 | 1
Shoulder operation (Injury, poisoning and procedural complications) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 0 | 1
Hemolytic anemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FSC + Tio (N=173) | Tiotropium (N=169)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 24 | 24
Headache (Nervous system disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.